CLINICAL TRIAL: NCT02648035
Title: Multicenter, Post-Marketing, Non-Interventional, Observational Study to Evaluate Persistence to Tocilizumab SC as Monotherapy or in Combination With cDMARD Treatment in RA Patients in Greece: the EMBRACE-SC Study.
Brief Title: EMBRACE-SC: Observational Study of Subcutaneous (SC) Tocilizumab Alone or in Combination With Conventional Disease-Modifying Antirheumatic Drugs (cDMARDs) in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29855
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subcutaneous Tocilizumab: Participants receiving treatment for rheumatoid arthritis (RA) with subcutaneous Tocilizumab alone or in combination with conventional disease-modifying antirheumatic drugs (DMARDs) according to approved label.
  Interventions: Biological: Tocilizumab

INTERVENTIONS:
Biological: Tocilizumab — Subcutaneous Tocilizumab according to approved label.
  Other Names: ACTEMRA

SUMMARY:
The purpose of this study is to evaluate the percentage of participants treated with subcutaneous (SC) Tocilizumab who are still on treatment after 52 weeks and the factors that play a major role in continuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

- Aged >/= 18 years of age with rheumatoid arthritis (RA) for whom the treating physician has made the decision to start subcutaneous (SC) Tocilizumab (TCZ) treatment according to approved label within 4 weeks prior to enrolment.

Exclusion Criteria:

* Participants who have been receiving Tocilizumab (TCZ) for more than 4 weeks prior to enrolment.
* Participants who have received TCZ in past treatments.
* Participants who have received treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational agent, whichever is longer) of starting treatment TCZ SC.
* Participants with a history of autoimmune disease or of any joint inflammatory disease other than rheumatoid arthritis (RA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with rheumatoid arthritis for whom the physician has made the decision to start subcutaneous Tocilizumab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09-22 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Still Receiving Subcutaneous Tocilizumab Therapy at 52 Weeks of Observation | At 52 weeks

SECONDARY OUTCOMES:
Health Assessment Questionnaire (HAQ) Score | At baseline, 24 and 52 weeks
Visual Analog Scale (VAS) Pain Score in a 100 mm Scale | At baseline, 24 and 52 weeks
Patient Global Assessment of Disease Activity (PtGA) Score in a 100 mm VAS Scale | At baseline, 24 and 52 weeks
Percentage of Participants with Clinically Significant Changes in Laboratory Values | At baseline, 24 and 52 weeks
Percentage of Participants on Subcutaneous Tocilizumab Alone Versus Combination Therapy | At baseline, 24 and 52 weeks
Percentage of Participants Involved in Subcutaneous Tocilizumab Patient Support Programs (PSPs) | At baseline, 24 and 52 weeks
Percentage of Participants with Adverse Events (AEs), including Serious Adverse Events (SAEs), Non-Serious Adverse Drug Reactions (nsADRs), Injection Site Reactions (ISRs), and Adverse Events of Special Interest (AESIs) | Up to 52 weeks
Percentage of Participants with Infections Events (IEs), Including Serious and Non-Serious IEs | Up to 52 weeks
Percentage of Participants with IEs with Laboratory Abnormalities | Up to 52 weeks
Percentage of Participants with Dose Modification of Methotrexate (MTX) or Other Non-Biologic Disease-Modifying Antirheumatic Drugs (DMARDs) Due to AEs or IEs | Up to 52 weeks
Percentage of Participants with Dose Modification of Subcutaneous Tocilizumab Due to AEs or IEs | Up to 52 weeks
Percentage of Participants on Glucocorticoids (GCs) with AEs | Up to 52 weeks
Disease Activity Score 28 (DAS28) | At baseline, 24 and 52 weeks
Percentage of Participants with Good/Moderate Response According to the Classification of the European League Against Rheumatism (EULAR) | At baseline, 24 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Greece (24):
  - Private Practice Rheumatology, Merantzis, Agrinio
  - Rheumatology Private Practice, Athens
  - General Hospital of Athens KAT, Rheumatology, Athens
  - Private Practice Rheumatology, Stavropoulos, Áno Patísia
  - Rheumatology Private Practice, Chania
  - Private Practice Rheumatology, Papadimitriou, Drama
  - Rheumatology Private Practice, Eleusina
  - ATTIKO Hospital_4th University Internal Medicine Clinic, Haidari
  - Private Practice Rheumatology, Georgiadis, Ioannina
  - Rheumatology Private Practice, Kalithea, Athens
  - Private Practice Rheumatology, Kotrotsios, Karditsa
  - General Hospital of Kavala; Rheumatology, Kavala
  - Rheumatology Private Practice, Kifissia
  - Private Practice Rehumatology, Ziogas, Larissa
  - General Hospital of Mytilini, Rheumatology, Mytilene
  - Private Practice Rheumatology, Trontzas, Néa Smýrni
  - Rheumatology Private Practice, Pátrai
  - Olympion Medical Center of Patras, Internal Medicine Clinic, Pátrai
  - Private Practice Rheumatology, Psaltis, Serres
  - Rheumatology Private Practice, Serres
  - Rheumatology Private Practice, Thessaloniki
  - General Hospital Agios Pavlos, Thessaloniki
  - Rheumatology Private Practice, Véroia
  - Rheumatology Private Practice, Volos